CLINICAL TRIAL: NCT07226180
Title: Beyond Genomics Functional Precision Oncology Research Study
Brief Title: Development and Application of Patient-Derived Models of Cancer
Status: Enrolling by invitation | Type: Observational
Sponsor: Certis Oncology Solutions, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: COS-IRB-001A - 220-23-CA
Record Dates: First submitted 2025-09-30; First posted 2025-11-10 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: solid tumor; PDX; patient-derived cancer models
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — biopsy or surgically obtained tumor tissue/fluid, blood specimens
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this observational study is to evaluate the clinical utility of investigational patient-derived cancer models, to assess the performance of biomarker-based therapeutic predictions in the patient-derived models.

Each participant in the observational study will have a piece of cancer removed as part of routine, physician direct care and grown in laboratory mice, where multiple anti-cancer drugs can be tested on it simultaneously. Additional data will be provided to the oncologist; interpretation of the results and any clinical actions are at the sole discretion of the oncologist.

DETAILED DESCRIPTION:
Participants are planned to undergo a procedure, such as a biopsy or surgery, as part of routine care. After enough tissue to complete all routine tests required for the participants' care are provided, if the participant decides to take part in this study, any leftover biopsy or surgically obtained tissue/fluid, and blood specimens will be sent to the Certis laboratory for testing. It will be required to provide details regarding the participants' biopsy, such as the date, location, and contact information for the study team performing the procedure. The oncologist will assist with this, and once confirmed, a kit will be sent to the location of the procedure to transport the specimen back to the Certis laboratory in San Diego, California.

The process of developing an individualized PDX (Patient Derived Xenograft) model is a 2-step process. The first is Initiation, where the biopsy is surgically implanted into 2-5 specialized research mice, depending on the size and quality of biopsy received, to allow it to grow. This identifies if the participants' tumor is suitable for growing in mice, as well as generating enough tumor material to conduct large studies on. This takes approximately 3-4 months.

The next step is Pharmacology. Here, selected tumors from the initial 5 mice are removed, dissected, and implanted into a larger number of mice, approximately 50. These mice are then divided into groups of 5, and each group is given a different anti-cancer therapy. Certis will work closely with the oncologist to select the therapies to test. The mice are treated for a period of 4 weeks, and the tumors are measured weekly to determine which therapies are better at treating the participants tumor in mice. The oncologist will be updated upon pre-specified study milestones.

ELIGIBILITY:
Inclusion Criteria:

* Solid tumor patients stage 2-4.
* Cancer patients who have been previously treated or shown resistance or refraction to standard-of-care therapies and where the implicated tissue has not been irradiated in the ten (10) weeks prior to excision.
* Patients with tumors are amenable to biopsy or surgery for fresh tissue and blood procurement as part of routine clinical care
* Patients must be referred by a healthcare professional
* Willingness for tissue samples used in future research
* Signed informed consent
* Willingness to share diagnosis, available genetic/molecular profiling data, treatment history, and treatment outcome monitoring

Exclusion Criteria:

* Failure to provide informed consent
* Inaccessible tumors for biopsy or unavailability of tumor tissue for research purposes
* Subjects under the age of 18
* Subjects with cognitive impairment
* Pregnant subjects
* Contraindications to undergoing a biopsy procedure
* No prior treatments, naive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of Hoag Memorial Hospital Presbyterian, Hoag Hospital Irvine, and Hoag Health Center Newport Beach
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-11-10 (Estimated); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
PDX Tumor Growth | 180 days
  The primary outcome of this study is the successful engraftment of patient-derived xenograft (PDX) tumors in the study animals. Engraftment success will be assessed by quantifying tumor growth using caliper measurements and/or magnetic resonance imaging (MRI). Successful engraftment will be defined as measurable and sustained tumor growth consistent with the characteristics of the original patient tumor.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Hoag Hospital Irvine, Irvine, California
  - Hoag Health Center Newport Beach, Newport Beach, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California

IPD SHARING:
Plan to Share IPD: No